CLINICAL TRIAL: NCT06482554
Title: Lumateperone for the Improvement of Apathy in Patients With Psychotic Symptoms.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Shawn McNeil, Principal Investigator, Louisiana State University Health Sciences Center Shreveport
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002212
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Apathy; Schizophrenia; Schizophrenia; Psychosis
Keywords: Schizophrenia; Schizoaffective; Psychosis; Psychotic
MeSH Terms: conditions — Lethargy; Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — lumateperone; Risperidone; Olanzapine; Quetiapine Fumarate; ziprasidone; Aripiprazole

STUDY DESIGN:
Intervention Model Description: Compare lumateperone treatment with existing medication
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumateperone (Active Comparator): 42mg capsule, once a day for 8 weeks
  Interventions: Drug: Lumateperone 42 mg
- Existing medication (Active Comparator): Existing medication reformulated in capsule, once or twice daily (as currently prescribed) for 8 weeks
  Interventions: Drug: Risperidone 2 mg

INTERVENTIONS:
Drug: Lumateperone 42 mg — Standard treatment with lumateperone
  Other Names: Lumateperone
  Arms: Lumateperone
Drug: Risperidone 2 mg — Standard treatment with other antipsychotic drugs
  Other Names: olanzapine; quetiapine; ziprasidone; aripiprazole
  Arms: Existing medication

SUMMARY:
This study is looking to determine if Lumateperone improves motivation in patients with schizophrenia or schizoaffective disorders who show high levels of apathy as judged by AES-C-Apathy (Apathy Evaluation Scale - Clinician - Apathy) assessment and to examine a possible correlation between improvement in apathy scores and changes in elements of the PANSS (Positive and Negative Syndrome Scale) due to treatment with Lumateperone.

DETAILED DESCRIPTION:
1. To determine if Lumateperone improves motivation in patients with schizophrenia or schizoaffective disorders who show high levels of apathy as judged by AES-C-Apathy assessment.
2. To examine a possible correlation between improvement in apathy scores and changes in elements of the PANSS (Positive and Negative Syndrome Scale) due to treatment with Lumateperone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18-65 that have been diagnosed with Schizophrenia, Schizoaffective Disorder or Schizophrenia Spectrum and Other Psychotic Disorders.
* A BPRS score > 35 at the screening visit.
* An AES-C score > 32 at the screening visit.
* If the subject is on a therapeutic regimen, that regimen must be stable for at least 30 days prior to screening. A therapeutic regimen may include medication, supplements, and/or probiotics.
* In the opinion of the Investigator, the subject is able to participate in all scheduled evaluations, and likely to be compliant and complete all required assessments.
* Female subjects of childbearing potential must not be pregnant or breast-feeding. Female subjects of childbearing potential must have a negative urine pregnancy test. Subjects of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control, which includes abstinence, while being treated on this study and for 30 days after the last dose of study drug.
* Must speak and understand English, as the consent and all evaluations will be conducted in English.
* Must be willing to take and pass a urine drug screen with a negative result in order to rule out psychotic symptoms due to drugs of abuse.

Exclusion Criteria:

* A BPRS score < 35 at the screening visit.
* An AES-C score < 32 at the screening visit.
* Have any clinically significant medical condition or an unstable intercurrent illness that would, in the opinion of the Investigator, preclude study participation.
* Are currently taking more than one antipsychotic medication.
* Are currently taking a long-acting injectable medication for psychotic symptoms.
* Have a substance use disorder or show a positive drug screen for stimulants.
* Are pregnant or of female sex with no evidence of measures for pregnancy prevention.
* Presence of dementia.
* Intellectual disability or cognitive impairment that would affect the symptom/apathy assessments, in the view of the investigator.
* A diagnosis of Parkinson's disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in AES-C Score | 8 weeks
  Difference between the mean change in the AES-C score from baseline (V1) to Week 8 (V3) for 42 mg/day lumateperone vs. current antipsychotic medication.

SECONDARY OUTCOMES:
Change in PANSS Score | 8 weeks
  Difference between the mean change in the PANSS score from baseline (V1) to Week 8 (V3) for 42 mg/day lumateperone vs. current antipsychotic medication.
Change in BPRS Score | 8 weeks
  Difference between the mean change in the BPRS (Brief Psychiatric Rating Scale) score from baseline (V1) to Week 8 (V3) for 42 mg/day lumateperone vs. current antipsychotic medication.
Correlations between AES-C and PANSS Scores | 8 weeks
  Correlation between the AES-C score at Week 8 (V3) and negative symptoms score from PANSS at Week 8 (V3) for 42 mg/day lumateperone in comparison to current antipsychotic medication.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn McNeil, MD, Principal Investigator — LSU Health Shreveport
Locations (1):
- LSU Health Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No